CLINICAL TRIAL: NCT06741267
Title: The Assessment of the Feasibility and Operational Performance of Automated System Bronchoscopy in a Simulated Environment: a Multicenter, Randomized-Controlled Trial.
Brief Title: The Assessment of the Feasibility and Operational Performance of Automated System Bronchoscopy in a Simulated Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Li Shiyue, Professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: automatic bronchoscopy
Record Dates: First submitted 2024-12-05; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-01

CONDITIONS: Compare Operational Performance of Three Technology in Lung Models

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RBS group (Other): physicians control robotic bronchoscopy system(RBS)
  Interventions: Device: RBS
- AB group (Other): physicians control automatic bronchoscopy(AB)
  Interventions: Device: AB
- ENB groups (Other): physicians control electromagnetic navigation bronchoscopy(ENB)
  Interventions: Device: ENB

INTERVENTIONS:
Device: RBS — physicians control RBS
  Arms: RBS group
Device: AB — physician control automatic bronchoscopy
  Arms: AB group
Device: ENB — physicians control electromagnetic bronchoscopy
  Arms: ENB groups

SUMMARY:
Recruit 30 trainee physicians from 6 centers and compare their performance in operating lung models using automatic bronchoscopy, robotic bronchoscopy, and electromagnetic navigation bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. The recruited participants were respiratory internal medicine trainees undergoing further training.
2. They were willing to undertake relevant training and complete the experiment persistently -

Exclusion Criteria:

If the participant has any previous clinical or simulated experiences involving electromagnetic navigation bronchoscopy, robotic bronchoscopy system, or fluoroscopy bronchoscopy, they will be excluded.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sampling time | During the bronchoscopy
  Sampling time , the time used to sample

SECONDARY OUTCOMES:
Total time | During the bronchoscopy
  total procedure time

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong 510163, Guangzhou, Guangdong, Chad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cold KM, Xie S, Nielsen AO, Clementsen PF, Konge L. Artificial Intelligence Improves Novices' Bronchoscopy Performance: A Randomized Controlled Trial in a Simulated Setting. Chest. 2024 Feb;165(2):405-413. doi: 10.1016/j.chest.2023.08.015. Epub 2023 Aug 23. PMID 37619664